CLINICAL TRIAL: NCT01962402
Title: Lorcaserin for Weight Loss Management in Patients on Antipsychotics: A Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Charles Nguyen, Psychiatrist, Southern California Institute for Research and Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VALB-1259
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lorcaserin with intensive diet counseling (Experimental): Patients will be taking lorcaserin 10mg tablet by mouth twice daily. In addition, patients will be provided with intensive dietary counseling to promote weight loss.
  Interventions: Drug: lorcaserin; Behavioral: Intensive dietary counseling

INTERVENTIONS:
Drug: lorcaserin — Patients will receive lorcaserin 10mg tablet, 1 tablet twice daily for 12 weeks.
  Other Names: Belviq
Behavioral: Intensive dietary counseling — All patients in the study will receive intensive dietary counseling, encouraging eating minimal carbohydrates and sugars.

SUMMARY:
The purpose of this study is to determine whether lorcaserin is effective for weight reduction in patients with weight gain as a result of antipsychotic medications.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients currently on atypical antipsychotics
* The patient's BMI is greater than or equal to 30 kg/m2 OR the patient's BMI is greater than or equal to 27 kg/m2 in the presence of at least one weight-related co-morbidity such as hypertension, type 2 diabetes mellitus, dyslipidemia, metabolic syndrome, obstructive sleep apnea, or degenerative joint disease such as osteoarthritis.
* Patient agreeable to follow up with provider at the scheduled appointments at week 1, week 2, week 4, week 8, week 12 and week 16 after initiation of medication.

EXCLUSION CRITERIA:

* Pregnancy in women or breastfeeding
* The patient has greater than mild aortic valve regurgitation, or moderate to greater mitral valve regurgitation
* Known hypersensitivity to lorcaserin
* The patient is taking another weight loss medication concurrently
* Dementia
* Age less than 18 or greater than 65
* No recent substance abuse within 3 months
* No suicidal ideation within 3 months
* Unable to give informed consent, unless patient is conserved, then the conservator can provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Weight loss | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
  The primary objective of this study is to evaluate the effectiveness of lorcaserin for weight loss management in patients on an antipsychotic agent. Will monitor the weight of the patient for evaluation.

SECONDARY OUTCOMES:
Evaluation of glucose control | At initial visit and at week 12 of the study
  Will evaluate lab values for fasting blood glucose, Hemoglobin A1c, and fasting insulin levels
Evaluation of cravings | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
  Using various questionnaires to evaluate cravings of various foods.
Monitoring of mood | At initial visit, then at week 4 and week 12 of the study
  Using standard questionnaires to evaluate mental health.
Evaluation of systolic blood pressure | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
Evaluation of diastolic blood pressure | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
Evaluation of pulse | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
Evaluation of body-mass index (BMI) | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
Evaluation of waist circumference | initial visit with provider, then at weeks 1, 2, 4, 8, 12, and 16 of the study
Evaluation of cholesterol control | At initial visit and at week 12 of the study
  Will measure fasting cholesterol labs, which will include total cholesterol, triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL)
Evaluation of electrolytes | At initial visit and at week 12 of the study
  Will monitor basic metabolic panel
Evaluation of liver | At initial visit and at week 12 of the study
  Will monitor liver enzymes
Evaluation of blood count | At initial visit and at week 12 of the study
  Will monitor blood count

CONTACTS AND LOCATIONS:
Locations (1):
- VA Long Beach, Long Beach, California, United States